CLINICAL TRIAL: NCT01291082
Title: Whole-body Magnetische Resonantie Voor Het Opsporen Van Bot- en Weke Delenmetastasen Bij patiënten Met Een Borstcarcinoom (MetaMaRBo)
Brief Title: Whole-body MR in Staging Bone and Soft Tissue Metastases in Breast Cancer Patients(MetaMaRBo)
Acronym: METAMARBO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Steven Pans, Medical Doctor radiologist, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S53057
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; metastasis; bone; diffusion MRI
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients: Breast cancer patients

SUMMARY:
Prospective MR-imaging study : role of magnetic resonance (MR) and Diffusion weighted imaging (DWI) MR in staging and therapy assessment in breast cancer patients with bone metastases.

DETAILED DESCRIPTION:
About 50 patients with a proven breast cancer and bone metastases will be included.

First step : staging

* nuclear bone scan
* Positron Emission Tomography (PET/CT)
* MR (whole body short tau inversion recovery (STIR)-sequence and T1-sequence and Diffusion weighted imaging (DWI),no contrast administration

Aim :

* Validation of whole body diffusion weighted imaging in detection of bone metastases and visceral metastases, comparing to Bone scan en PET/CT results.
* To calculate cut-off values for DWI for bone and visceral metastases.

Second step : therapy follow-up/therapy assessment.

* Two groups of patients (oncologist takes the decision about therapy)

  1. Patients treated by chemotherapy
  2. Patients treated by hormonal therapy
* on week 3, 12-16 and 52 in the chemotherapy or hormonal therapy-setting, a whole body MR (same protocol, no contrast) will be performed.

End-point:

Whole body MR with DWI is useful and reliable to assess the treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a proven breast cancer (by biopsy or imaging)
2. Bone metastases proven by MR, PET-CT or Bone. Patients with visceral metastases can be included if bone metastases are also present.
3. Patient with an informed consent.

Exclusion Criteria:

1. Patients with a single bone metastasis treated by Radiotherapy will be excluded.
2. Patients with contra-indication for MRI: pacemaker, cochlear implant, non MR compatible devices (Baclofenpump).
3. Claustrophobia
4. Patient in a bad general condition.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Validation of whole body diffusion weighted MRI in breastcancer patients | 6 months
  whole body MRI will be correlated to the nucleair bone scan and PET-CT

SECONDARY OUTCOMES:
Whole body MRI with diffusion weighted imaging is a reliable imaging tool for therapy assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pans, MD, Principal Investigator — UZ Leuven Dept Radiology
Locations (1):
- University Hospitals Leuven, Leuven, Belgium